CLINICAL TRIAL: NCT03456089
Title: Measurement of Bladder Pressure With a Novel External Device, Comparison to Urodynamics Testing
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Cooper (Other)
Responsible Party: Sponsor-Investigator, Christopher Cooper, Associate Dean, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201702822
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Urinary Bladder, Neurogenic; Urodynamics
Keywords: urodynamics; neurogenic; bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neurogenic Bladder Patients (Other): Patients with neurogenic bladder undergoing urodynamics testing
  Interventions: Diagnostic Test: Urodynamics Testing

INTERVENTIONS:
Diagnostic Test: Urodynamics Testing — Urodynamics utilizes a small catheter to fill the bladder and continuously measure pressure and volume giving information on bladder function and compliance

SUMMARY:
The investigators have developed a novel pressure monitoring device that hooks to standard urinary catheters. The investigators will be testing how the pressure measurements recorded with this device compare to the gold standard measurement of urodynamics.

DETAILED DESCRIPTION:
For patients with neurogenic bladder, regular monitoring of bladder pressure and capacity is a critical component of maintaining renal and urinary health. This monitoring is currently done by in-office urodynamics testing (UDS). This testing is done intermittently, leaving open the possibility of worsening of bladder function and renal deterioration between testing sessions.

This study utilizes a novel pressure monitoring device which is portable and hooks to the end of a standard urinary catheter. The investigators will be investigating if this device can achieve similar pressure measurements as UDS. The investigators hope is that this device will provide similar measurements to UDS, and can be developed as a home bladder-pressure monitoring tool.

This study will enroll children with neurogenic bladder who are currently undergoing UDS as part of their regular care. The measurements will be taken as part of the standard UDS protocol (with insertion of the UDS catheter) and will then be compared to the values obtained with UDS testing.

ELIGIBILITY:
Inclusion Criteria:

* must have diagnosed neurogenic bladder
* undergoing urodynamics testing as part of routine clinical care

Exclusion Criteria:

-None

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Bladder Pressure | During UDS testing
  Pressure of the bladder at bladder capacity

CONTACTS AND LOCATIONS:
Overall Officials: Chris Cooper, MD, Principal Investigator — MD
Locations (1):
- University of Iowa Hospitals and Clinics, Department of Urology, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No